CLINICAL TRIAL: NCT06294860
Title: Evaluation of Biological Age in Children With GH Deficiency Undergoing Hormone
Brief Title: Biological Age in Children With GH Deficiency Undergoing Hormone Replacement Therapy
Acronym: ETABIOGHD
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C317
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Growth Hormone Deficiency; Short Stature
Keywords: Growth hormone deficiency; Replacement therapy; Recombinant growth hormone; Short stature; Biological age; Epigenetic
MeSH Terms: conditions — Dwarfism, Pituitary; Dwarfism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — From the leucocytes isolated from the samples taken at T0 and T6, the DNA is extracted. The DNA methylation is performed with sodium bisulfite and PCR- Pyrosequencing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hormone replacement therapy with rhGH: Each subject will be treated with hormone replacement therapy with rhGH with a dose of 0.025-0.035 mg/kg body weight per day (or 0.7-1.0 mg/ m2 body surface area per day) for a period of 6 months.

SUMMARY:
The primary objective of the study is to evaluate the epigenetic age in children with GH deficiency, before and after 6 months of treatment with growth hormone replacement therapy. The secondary objective is to correlate the epigenetic age with the auxometric and biochemical parameters used in the clinical-endocrinological practice. The results of the study will be useful to set up the clinical and biochemical follow-up of the hormone replacement therapy with rhGH and to understand the biomolecular mechanisms at the base of the debated "anti" or "pro" aging action of GH, the most important anabolic hormone of the human organism.

DETAILED DESCRIPTION:
12 children of both sexes affected by an isolated GH deficiency (defined according to the criteria provided by the note 39 AIFA for this pathology: short stature: ≤ -3 DS or ≤ -2 DS; growth rate/year ≤ -1.0 DS per age and sex evaluated at a distance of at least six months; GH peak at two different pharmacological stimulation tests < 8 ng/ml), recruited at the Regional Reference Centre for Growth Disorders, Istituto Auxologico Italiano, IRCCS, Milano. The exclusion criteria for the study (and from the rhGH treatment) are the presence of organic hypothalamic-pituitary pathologies (diagnosed through encephalic RMN).

In basal conditions (pre-treatment), the clinical and anthropometric/auxometric data (height, weight, BMI) are collected, including the evaluation of the body composition with bioelectrical impedance analysis. The same evaluations is repeated after 6 months of treatment with recombinant growth hormone (see below).

Each subject is treated with replacement therapy with rhGH at a dose of 0.025-0.035 mg/kg body weight per day (or 0.7-1.0 mg/ m2 body surface area per day).

Blood samples for the determination of: glycemia, insulin, HbA1C, triglycerides, total cholesterol, LDL, HDL, hsPCR, IGF-1, osteocalcin, ICTP, and PIIINP are collected at T0 (before the start of the hormone replacement therapy with rhGH) and at T6 (after 6 months of rhGH, approximately 10-12 from the last dosing).

From the leucocytes isolated from the samples taken at T0 and T6, the DNA is extracted. The DNA methylation is performed with sodium bisulfite and PCR- Pyrosequencing.

The biological age (epigenetic) is measured with two algorithms of Zbiec-Piekarska and of Daunay, based on DNA methylation level in specific loci. To have an estimate of the epigenetic age (biological) that is independent of the chronological age, a defined measure defined as age acceleration will be used, for which calculation a linear regression model will be applied with the chronological age as independent variable and the epigenetic age as dependent variable; the difference between the observed value and the predicted value from the model represents the age acceleration due to a properly epigenetic effect. In case the epigenetic age is higher than the chronological age, the age acceleration has a positive value expressed in years, otherwise negative.

ELIGIBILITY:
Inclusion Criteria:

* children of both sexes
* age 5-15 years affected by isolated GH deficiency according to the criteria provided by note 39 AIFA for this pathology (short stature: ≤ -3 DS or ≤ -2 DS; growth rate/year ≤ -1.0 DS per age and sex evaluated at a distance of at least six months; GH peak at two different pharmacological stimulation tests < 8 ng/ml).

Exclusion Criteria:

- presence of organic hypothalamic-pituitary pathologies (diagnosed through encephalic NMR).

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with isolated growth hormone deficiency
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Measurement of biological (epigenetic) age | Baseline and after 6 months of substitutive treatment with recombinant growth hormone
  The biological age (epigenetic) is measured in basal condition (T0) and after 6 months of treatment with recombinant growth hormone with two algorithms (Zbiec-Piekarska and Daunay), based on DNA methylation level in specific loci. To have an estimate of the epigenetic age (biological) that is independent of the chronological age, we use age acceleration, for whose calculation we apply a linear regression model with the chronological age as independent variable and the epigenetic age as dependent variable; the difference between the observed value and the predicted value from the model is the age acceleration due to a properly epigenetic effect. In case the epigenetic age is higher than the chronological age, the age acceleration has a positive value expressed in years, otherwise negative.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Sartorio, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy